CLINICAL TRIAL: NCT00246298
Title: A Randomized, Open-Label Study Assessing the Efficacy of Initiating PROCRIT (Epoetin Alfa) Dosing at Q2W vs. PROCRIT Dosing at QW in Anemic HIV-infected Subjects
Brief Title: A Study to Assess the Effectiveness of PROCRIT (Epoetin Alfa) Dosing Every 2 Weeks Versus Once a Week in Anemic HIV-infected Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: OBI business decision not to complete any additional research in HIV.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR003220
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-03

CONDITIONS: Anemia; HIV
Keywords: Anemia; erythropoetin; Epoetin alfa; erythropoietin recombinant; HIV infection; HIV; AIDS
MeSH Terms: conditions — Anemia; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to determine if PROCRITÂ® (a glycoprotein that stimulates red blood cell production) initiated at once every 2 weeks dosing is as effective as PROCRITÂ® initiated at once a week dosing, in increasing hemoglobin levels in anemic HIV-infected subjects.

DETAILED DESCRIPTION:
In the Highly Active Antiretroviral Treatment (HAART) era, anemia is one of the most common abnormalities in HIV-infected subjects. Epoetin alfa is proven to increase hemoglobin levels and improve quality of life in HIV-infected subjects. Although there are data to show that epoetin alfa dosed weekly significantly increases hemoglobin to a target level of 13 g/dL and every other week dosing can maintain target hemoglobin, there is no data to show that initiation of epoetin alfa every 2 weeks will increase hemoglobin levels significantly.

This randomized, two-arm, open-label study will evaluate if initiating PROCRIT® every other week dosing is as effective as initiating PROCRIT® weekly dosing, in increasing hemoglobin in anemic HIV-infected subjects. The Screening phase will start 2 weeks prior to the first dose of PROCRIT®. HIV-infected subjects who have a hemoglobin level of <12.0 g/dL and are on a stable antiretroviral regimen will be screened for study eligibility. In the treatment phase, subjects will be randomized in a 1:1 ratio to receive 40,000 IU PROCRIT® subcutaneous injections either weekly (QW) or every other week (Q2W). The primary endpoint is the change in hemoglobin from baseline to the end of study at Week 12. The safety and tolerability of PROCRIT® in this subject population will be assessed by evaluating adverse events, laboratory results and vital signs. The total duration of this study is 14 weeks, including a 2-week screening phase and a 12-week treatment phase. The primary hypothesis is that the mean increase in hemoglobin for subjects receiving PROCRIT® every 2 weeks is not lower than those receiving weekly PROCRIT® dosing by more than 1 g/dL. Subjects will initially receive 40,000 IU PROCRIT® subcutaneous injections either weekly (QW) or every other week (Q2W), with subsequent dose adjustments, if appropriate. The maximum length of PROCRIT® treatment for this study is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be documented HIV positive and on a stable antiretroviral regimen for at least four weeks prior to enrollment
* have a hemoglobin level <12.0 g/dL
* have not undergone cancer therapy (chemotherapy and/or radiation therapy) within 12 months prior to enrollment

Exclusion Criteria:

* History of acute, symptomatic opportunistic infection or other acute AIDS defining illness within six months of enrollment
* History of any primary hematologic disease
* Have anemia attributable to factors other than HIV infection (i.e. iron, or vitamin B12 deficiency, hemolysis, or gastrointestinal bleeding)
* Have Hepatitis C virus (HCV) co-infection
* Have uncontrolled or severe cardiovascular disease including recent myocardial infarction, hypertension, or congestive heart failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-10; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin from baseline to the end of study at Week 12

SECONDARY OUTCOMES:
Safety and tolerability of every other week dosing and once a week dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Randomized, Open Label Study Assessing the Efficacy of Initiating PROCRIT Dosing at Q2W vs. PROCRIT Dosing at QW in Anemic HIV-infected Patients — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=511&filename=CR003220_CSR.pdf